CLINICAL TRIAL: NCT01914276
Title: A Pilot Study of Postoperative Lower-extremity Lymphedema and Quality of Life Among Women Undergoing Endometrial Cancer Staging Surgery
Brief Title: Lymphedema in Endometrial Cancer
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00047483
Record Dates: First submitted 2013-07-31; First posted 2013-08-02 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Lower Extremity Lymphedema; Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Objectives: (1) To determine the incidence of lower-extremity lymphedema after staging surgery for endometrial cancer; (2) to describe lymphedema-related morbidity after staging surgery for endometrial cancer and (3) to evaluate pre- and post-operative quality of life in women with endometrial cancer who undergo staging surgery.

Data analysis and risk/safety issues: The proposed study will consist of a convenience sample of women who undergo minimally invasive surgery for endometrial cancer over a 1 year period. The investigators anticipate enrollment of 75 to 100 women. Frequency tables and difference with its 95% exact confidence intervals between pre-and post-operative lower extremity lymphedema measurements and quality of life questionnaires will be estimated.

ELIGIBILITY:
Inclusion Criteria:

1. women older than 18 years old,
2. endometrial cancer,
3. suitable candidates for surgery,
4. scheduled to undergo laparoscopy or robotic-assisted (RA) laparoscopy for endometrial cancer at Duke University Medical Center (DUMC),
5. no severe physical or mental comorbidity

Exclusion Criteria:

1. metastatic disease,
2. laparotomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: (1) women older than 18 years old, (2) endometrial cancer, (3) suitable candidates for surgery, (4) scheduled to undergo laparoscopy or robotic-assisted (RA) laparoscopy for endometrial cancer at Duke University Medical Center (DUMC), (5) no severe physical or mental comorbidity
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-10; Primary Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
change in incidence of lower-extremity lymphedema | 1 month, 6-9 months and 12-18 months after staging surgery for endometrial cancer

SECONDARY OUTCOMES:
change in lymphedema-related morbidity | 1 month 6-9 months and 12-18 months after staging surgery for endometrial cancer

OTHER OUTCOMES:
change in quality of life in women with endometrial cancer who undergo staging surgery | pre-operatively, 1 month post-op, 6-9 months and 12-18 months post-op
  The study team plans to measure QoL via 2 questionnaires, specifically the EQ-5D and FACT-G. FACT-G and EQ-5D-derived utility scores will be calculated and summarized pre- and post-operatively for all patients using descriptive statistics (means, medians, ranges). The difference with 95% exact confidence intervals between pre- and post-operative FACT-G scores and EQ-5D utility scores obtained at each post-operative visit (t1, t2, & t3) will be estimated.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Havrilesky, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States